CLINICAL TRIAL: NCT03207646
Title: Smartphone GUIded MeDication AdherencE and Rehabilitation in Patients With Coronary Artery Disease (smartGUIDE)
Brief Title: Smartphone GUIded MeDication AdherencE and Rehabilitation in Patients With Coronary Artery Disease
Acronym: smartGUIDE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The company that provided the intervention shut down & withdrew the intervention
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Mintu Turakhia, Associate Professor of Cardiovascular Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 39555
Record Dates: First submitted 2017-06-16; First posted 2017-07-05 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Coronary Artery Disease; Acute Coronary Syndrome
Keywords: Cardiac Rehabiliation; Percutaneous Coronary Intervention; Cardiovascular Risk Factor; Digital Health Solution; Medication Adherence
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome; Medication Adherence

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to either the experimental arm or the 'no intervention' (control) arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- smartphone-based cardiac rehabilitation (Experimental): The BrightHeart® mobile application is installed on the smartphone and a heart coach set up and guides the participant through a cardiac care program.
  Interventions: Other: BrightHeart®
- Control (No Intervention): Standard-of-care alone.

INTERVENTIONS:
Other: BrightHeart® — BrightHeart® has two components: smartphone mobile based application and a human coach. It is a combined approach of medication adherence, exercise, diet, sleep and stress reduction.
  Arms: smartphone-based cardiac rehabilitation

SUMMARY:
This study evaluates a smartphone-based cardiac rehabilitation program in adults with coronary artery disease. Half of patients will participate in a smartphone-based cardiac rehabilitation program while the other half will receive standard-of-care.

DETAILED DESCRIPTION:
Cardiac rehabilitation as a means to improve lifestyle-based risk factor modification, remains poorly prescribed and utilized, often due to the lack of access to programs, poor insurance coverage, cost, or patient or physician motivational factors. Low-cost solutions that can improve patient adherence to medications, risk factor reduction, and exercise could improve cardiovascular outcomes and cost-effectiveness compared to current care models.

ELIGIBILITY:
Inclusion criteria:

I. ≥ 18 years of age

II. Patient at Stanford Health Care with evidence of CAD (atherosclerosis of one or more coronary arteries or clinical evidence or documentation of ischemia, infarction) OR a diagnosis related to CAD (i.e. ischemic heart disease ICD-10-Code: I20-25).

III. Prescription of a P2Y12 antagonist and/or a statin for an anticipated duration of at least 3 months following discharge

IV. Possession of a compatible (iPhone 5s or later; OS 8.1 or higher) smartphone with an active phone number and data plan. The smartphone must be in continued possession of the participant. It may not be a shared device and must exclusively remain in the possession of the participant during the study period. The smartphone must have an active cellular phone number and cellular data subscription. Wi-Fi internet capability is not a substitute for an active cellular data plan.

V. Must sign an informed consent form (ICF) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study.

VI. Willing to have the mobile application installed on a smartphone and use it every day during the entire study period VII. Willing to provide oral confirmation indicating that he/she is currently not using a medication adherence application.

VIII. Ability to read and understand English.

Exclusion criteria:

Any potential participant who meets any of the following criteria will be excluded from participating in the study:

I. Anticipated inability to adhere to the mobile application (BrightHeart®) based on opinion of site Principal Investigator (PI).

II. Current use of adherence tracking devices, electronic, smartphone or computer applications, including but not limited to smart pill bottles, pill timers, radiofrequency tagged medications or dispensers, mobile applications, or automated phone reminders. Pill organizers that remind participants when to take medicine with beeps or alerts are exclusion.

a. Note: Pharmacy and health care plan automated refill reminders are permitted and are not exclusion. Pill organizers or containers that only compartmentalize a participant's medications based on days of the week are not exclusion.

III. Cognitive, visual, hearing, voice, or motor impairment that would prevent completion of study procedures or use of mobile phone. Co-morbidities that would preclude participation (e.g. ongoing chemotherapy) or planned hospitalization for complex procedures as determined by the PI (e.g. bypass, valve or aortic surgery, transarterial valve replacement) IV. End-stage of one of the following: heart failure (using left ventricular assist device or listed for heart transplantation), renal disease, lung disease, liver disease.

V. Any condition with a life expectancy less than 3 months. VI. Employee of the investigator or study site, with direct involvement in the proposed study or other studies under the direction of that investigator or study site, as well as family members of the employees or the investigator VII. Any other condition as determined by the PI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2018-05-09 (Actual); Study Completion 2018-08-17 (Actual)

PRIMARY OUTCOMES:
Medication adherence | Baseline through End of Study visit - approximately 90 days per participant.
  The proportion of days coverd (PDC) expressed as a percentage but considered as a continuous variable of the composite of the prescribed P2Y12 receptor antagonist and/or the statin.

SECONDARY OUTCOMES:
Medication adherence II | Baseline through End of Study visit - approximately 90 days per participant.
  Proportion of participants with PDC ≥ 80% of the composite of the P2Y12 receptor antagonist and/or the statin
Medication adherence III | Baseline through End of Study visit - approximately 90 days per participant.
  The PDC of each medication of the composite
Medication adherence IV | Baseline through End of Study visit - approximately 90 days per participant.
  Proportion of participants with PDC ≥ 80% of each of the composite
Medication adherence V | Baseline through End of Study visit - approximately 90 days per participant.
  Mean time from discharge to first fill
Medication persistence | Baseline through End of Study visit - approximately 90 days per participant.
  proportion of patients with an active prescription at three months of a statin and P2Y12 inhibitor
Cardiovascular risk factors I | Baseline through End of Study visit - approximately 90 days per participant.
  Serum LDL-C at End of Study
Cardiovascular risk factors II | Baseline through End of Study visit - approximately 90 days per participant.
  Proportion of participants within target blood pressure (<140/90 mmHg or <130/80 mmHg for patients with diabetes mellitus or chronic kidney disease) at End of Study
Cardiovascular risk factors III | Baseline through End of Study visit - approximately 90 days per participant.
  Proportion of participants with HbA1c ≤ 7% at End of Study (only if diabetes mellitus was known at time of inclusion)
Cardiovascular risk factors IV | Baseline through End of Study visit - approximately 90 days per participant.
  Change in body weight from baseline to End of Study
Cardiovascular risk factors V | Baseline through End of Study visit - approximately 90 days per participant.
  Change in quality of life (measured by EQ-5D-3L14) from day 3-10 after discharge to End of Study
Cardiovascular risk factors VI | Baseline through End of Study visit - approximately 90 days per participant.
  Change in patient activation (measured by PAM®1015) from day 3-10 after discharge to End of Study
Cardiovascular risk factors VII | Baseline through End of Study visit - approximately 90 days per participant.
  Physical activity at End of Study (measured by a physical acitivity questionnaire)
Exploratory I: Rehospitalization | Baseline through End of Study visit - approximately 90 days per participant.
  30-day rehospitalization for any reason
Exploratory II: Cardiovascular outcomes | Baseline through End of Study visit - approximately 90 days per participant.
  Major adverse cardiac events (MACE) defined as: Death, myocardial infarction, acute coronary syndrome, out of hospital cardiac arrest, stent thrombosis, repeat revascularization at 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Minang (Mintu) Turakhia, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Healthcare, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No